CLINICAL TRIAL: NCT06805604
Title: Clinical Performance and Patients Satisfaction of Innovative Digital Techniques for Fabrication of Monolithic Ceramic Crowns
Brief Title: Digital Techniques
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Eman Hafez Elfky, assistant lecturer, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P-CR-23-15
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-09

CONDITIONS: Monolithic Ceramic Crowns Fabricated by Different Digital Techniques
Keywords: digital techniques

STUDY DESIGN:
Intervention Model Description: study is performed on 3 groups
  - Different digital techniques used for fabrication of the monolithic ceramic crowns were chosen for the current study; milled zirconia for the group (I) and milled hybrid for the group (II) and 3D-printed hybrid for the group (III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- milled zirconia crowns (Experimental): this group was received milled zirconia crowns on their posterior molars indicated for full coverage restorations.
  Interventions: Procedure: Each group was received monolithic ceramic crowns fabricated using different technique
- milled hybrid ceramic crowns (Experimental): this group was received milled hybrid ceramic crowns on their posterior molars indicated for full coverage restorations.
  Interventions: Procedure: Each group was received monolithic ceramic crowns fabricated using different technique
- 3d printed hybrid ceramic crowns (Experimental): this group was received 3d printed hybrid ceramic crowns on their posterior molars indicated for full coverage restorations.
  Interventions: Procedure: Each group was received monolithic ceramic crowns fabricated using different technique

INTERVENTIONS:
Procedure: Each group was received monolithic ceramic crowns fabricated using different technique — -Different digital techniques used for fabrication of the monolithic ceramic crowns were chosen for the current study, Clinical performance of all crowns regarding; marginal adaptation, fracture of restoration during service, color stability and wear behavior will be evaluated according to Modified United States Public Health Service (USPHS) Criteria at base line (1 week), 3 and 6 months after cementation of crowns.

SUMMARY:
The present study is performed to evaluate clinical performance and patient satisfaction of innovative digital techniques for fabrication of monolithic ceramic crowns

DETAILED DESCRIPTION:
Digital dentistry has progressed rapidly in the last few years, primarily to improve and enhance the practice of dentistry through the advancement in digital tools and techniques, providing improved accuracy and precision, enhancing patient experience, increasing efficiency and productivity, thereby resulting in better treatment outcomes, whilst also improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with posterior molars indicated for full coverage restorations.
* Patient able to physically and psychologically tolerate conventional restorative procedures.

Exclusion Criteria:

* Patient in the growth stage with partially erupted teeth.
* Patient with poor oral hygiene and motivation.
* Patients with parafunctional habits.

Ages: 21 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
the clinical performance, color stability and wear behavior of monolithic ceramic crowns fabricated using innovative digital techniques. | baseline, 3months and 6 months after crown cementation
  Clinical performance of all crowns regarding; marginal adaptation, fracture of restoration during service, color stability and wear behavior will be evaluated according to Modified United States Public Health Service (USPHS) Criteria at base line (1 week), 3 and 6 months after cementation of crowns.
  * Color stability will be evaluated using a spectrophotometer.
  * Wear of restorations will be evaluated using a software analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dental medicine for girls Al-Azhar university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diken Turksayar AA, Demirel M, Donmez MB, Olcay EO, Eyuboglu TF, Ozcan M. Comparison of wear and fracture resistance of additively and subtractively manufactured screw-retained, implant-supported crowns. J Prosthet Dent. 2024 Jul;132(1):154-164. doi: 10.1016/j.prosdent.2023.06.017. Epub 2023 Jul 20. PMID 37479623